CLINICAL TRIAL: NCT06331780
Title: Refractive Status and Accommodation Response Under Different Experimental Conditions.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: WS10370; 2023-A02153-42 (Other: ANSM (France))
Record Dates: First submitted 2024-03-12; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Accommodation Disorder; Accommodative Fatigue; Accommodative Inertia
MeSH Terms: interventions — Visual Acuity; Coping Inventory for Stressful Situations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Closed-field Aberrometer (Experimental): Objective refraction at different distances with Shack-Hartmann Aberrometer
  Interventions: Device: Visual acuity; Device: Objective refraction; Device: Objective monocular accommodation amplitude measurement; Device: Subjective monocular accommodation amplitude measurement with the "Push-Up" method; Device: Subjective monocular accommodation facility measurement with the "Rock" method:; Other: CISS Questionnaire; Other: Difficulty assessment questionnaire; Other: Subjective evaluation questionnaire

INTERVENTIONS:
Device: Visual acuity — VA will be measured with an Early Treatment Diabetic Retinopathy Study (ETDRS) chart
Device: Objective refraction — Objective refraction will be measured using an auto-kerato-refractometer/aberrometer
Device: Objective monocular accommodation amplitude measurement — Objective monocular accommodation amplitude measurements are obtained dynamically by measuring the subject's dioptric change while the participant focuses on a virtual object that moves from distance
Device: Subjective monocular accommodation amplitude measurement with the "Push-Up" method — The subjective monocular accommodation amplitude measurements are carried out by the "push-up" method and proceeds as follows:
  * The ECP presents a near vision test card corresponding to a 0.8 (8/10) acuity line, or the smallest readable line if acuity is poor, or the smallest readable text.
  * Instructions to the subject: "Look at the smallest line of letters and try to see them clearly for as long as possible when I bring them closer; tell me when they start to blur and stay blurred.
  * The ECP slowly brings the test card closer
  * The ECP note the distance of the test card from the glasses as soon as the vision is blurred. Continue to move the test closer to check that vision remains blurred.
  The amount of accommodation in this eye is equal to the proximity (= 1/distance) of the test when the blur is just perceived.
Device: Subjective monocular accommodation facility measurement with the "Rock" method: — The subjective monocular accommodation facility measurements are carried out by the "Rock" method and proceeds as follows:
  * The ECP presents at 40cm a near vision test card corresponding to 80% of the VA.
  * The ECP gives to the participant a flipper +/- 2 Dioptre
  * Instructions to the subject: "Look at the test" and add the -2.00 D (Sphere) flipper, as soon as it's clear, return the flipper to present a +2.00 D (Sphere), as soon as it's clear, return the flipper etc… You have to do the maximum number of rotations in one minute.
Other: CISS Questionnaire — This questionnaire relating to the use of the near vision will be submitted
Other: Difficulty assessment questionnaire — After each near vision measurement, the participant should rate, on a Visual Analogic Score (0-10), the difficulty encountered, from 0: extremely easy to 10: extremely difficult. The participant may also specify the reasons for the difficulty(ies) encountered during the measurement.
Other: Subjective evaluation questionnaire — A subjective evaluation questionnaire will be submitted to the participants at the end of the visit.

SUMMARY:
Eye Care Professionals (ECPs) massively use auto-refractors during the patient journey to measure the objective refractive error: starting point of the subjective eye refraction. These devices provide objective information about the refractive and accommodative state of the eye, useful for the ECP to perform a complete eyesight test. Auto-refractor data for the distance vision are repeatable and accurate but near vision information are not enough reliable to build an accurate near vision routine exam. Previous internal studies, with auto refractors currently on the market, have shown that, during accommodation measurements, a large proportion of participants had a lower accommodative response than expected.

DETAILED DESCRIPTION:
Clinical Development stage and rationale

The clinical development stage is pilot stage as defined in ISO 14155:2020 (Annex I section 1.3.2).This clinical investigation is an exploratory clinical investigation as mentioned in the Medical Device Regulation EU 745/2017, also named early feasibility clinical investigation in the ISO 14155:2020. The necessity of such clinical investigations is more precisely described by the Food and Drug Administration (FDA) (Attachment E CDRH Final Guidance Cover Sheet) and Agence Nationale de Sécurité du Médicament et des produits de santé (ANSM), where they detail the importance of exploratory studies in pivotal investigation design.

Medical devices often undergo design improvement during development, with refinement during lifecycles beginning with early research, extending through investigational use and initial marketing of the approved or cleared product, and continuing to subsequently approved or cleared commercial device versions.

Objectives and hypotheses of the clinical investigation

This clinical investigation explores new ways of measuring accommodative response, particularly regarding the dynamics and amplitude of response: we chose to vary several parameters.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer: man or woman from 18 to 40 years old,
* Subject declares that his last visit to an ophthalmologist was less than 12 months ago,
* Subjects without a reported pathology, deficit or disorder that can interfere with visual or cognitive functions,
* Subjects, healthy volunteers who have been fully informed of the investigation and signed the informed consent form of the investigation,
* Subjects available for the investigation visits (at least 2 hours),
* Subjects able to appoint a visit in the investigator's site,
* Subjects able to read and understand the protocol (in French), follow the instructions, and give their informed consent approval.

Exclusion Criteria:

* Subjects with spherical equivalent wearing compensation (or fully compensate by contact lenses) ranging out from -3.00 to + 3.00 Dioptres in both eyes,
* Subjects with an astigmatism wearing compensation (or fully compensate by contact lenses) more than 1.00 Dioptres (>1,00DC) in both eyes,
* Subjects with a best compensated monocular VA < 8/10 (>0.1logMAR),
* Persons subject to a legal protection measure (guardianship, curatorship, safeguard of justice, etc.) or unable to express their consent (see Article L 1121-8 of the CSP)
* Persons deprived of their liberty by judicial or administrative decision and persons hospitalised without their consent (article L1121-6 of the CSP),
* Subjects under exclusion period from another investigation,
* Women pregnant or breastfeeding; (Article L1121-5),
* Subjects with a reported neurologic disorder, particularly epileptic or sensory motor troubles,
* Subjects with implanted electronic medical device such as (pacemaker or hearing aid),
* Subjects with a reported severe ocular disease leading to a visual field decrease, VA deficiency or glare sensitivity,
* Subjects with monophtalmia
* Subjects who had ocular surgeries (including aphakia or pseudophakia (intraocular lenses), refractive surgery or trauma),
* Subjects who are ESSILOR INTERNATIONAL employees
* Subjects who are not affiliated to a social security scheme or are beneficiaries of such a scheme (article L1121-8-1 of the CSP).
* Subject with fixation disorder: impossibility to maintain fixation on visual target.
* Subjects who cannot stay comfortable during the tests (e.g. with neck pain ...).
* Pupil abnormality (unusual shape, size <3mm)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Accommodative response measured with closed-field aberrometer with different target displacement methods | One day (measurements are taken during the single visit)
  Accommodative response (Dioptries)
Accommodative response measured with closed-field aberrometer with different displayed targets | One day (measurements are taken during the single visit)
  Accommodative response (Dioptries)
Objective refraction measured with closed-field aberrometer and two camera exposure times | One day (measurements are taken during the single visit)
  Sphere (Dioptries), Cylinder (Dioptries), Axis (°) and High Order Aberrations (Zernike polynomials)

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme Gillet, Principal Investigator — ESSILOR INTERNATIONAL - Division Instruments
Locations (1):
- Essilor International - Ci&T 2, Créteil, France